CLINICAL TRIAL: NCT01742832
Title: Double-Blind Switch Study of Vilazodone in the Treatment of Major Depressive Disorder Following Partial Response to or Inability to Tolerate a Generic SSRI
Brief Title: Double-Blind Treatment of Major Depressive Disorder With Vilazodone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012MDDVilaz
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Major Depressive Disorder
Keywords: Vilazodone; Citalopram; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vilazodone Hydrochloride; Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vilazodone (Active Comparator): A fixed dose titration (with doses ranging from 10mg to 40mg/day) will be used. Subjects will take 10mg/day for 1 week, 20mg/day for 1 week and then 40mg/day.
  Interventions: Drug: Vilazodone
- Citalopram (Placebo Comparator): For those assigned to citalopram, the dose of citalopram will be maximized to 40mg/day. For those assigned to vilazodone, their citalopram dose will be maintained at 20mg/day for 1 week, then reduced to 10mg/day for 1 week, then switched to vilazodone 10mg/day.
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Vilazodone — A fixed dose titration (with doses ranging from 10mg to 40mg/day) will be used. Subjects will take 10mg/day for 1 week, 20mg/day for 1 week and then 40mg/day.
  Arms: Vilazodone
Drug: Citalopram — For those assigned to citalopram, the dose of citalopram will be maximized to 40mg/day. For those assigned to vilazodone, their citalopram dose will be maintained at 20mg/day for 1 week, then reduced to 10mg/day for 1 week, then switched to vilazodone 10mg/day.
  Arms: Citalopram

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of vilazodone for the treatment of major depressive disorder versus citalopram. Doctors want to determine if vilazodone is effective for the treatment of major depressive disorder in those who have not responded to generic selective serotonin reuptake inhibitors (SSRI), which is a class of anti-depressant drugs such as Prozac, Lexapro, Paxil, or Zoloft. Both vilazodone and citalopram have been approved for the treatment of major depressive disorder. This research is being done because the researchers want to find out if vilazodone works in reducing the symptoms of depression significantly more than a generic SSRI.

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the efficacy and safety of switching to Vilazodone in patients with major depressive disorder (MDD) who are unresponsive to, only partially responsive to, or cannot tolerate a trial of the generic SSRI, citalopram (e.g., "partially responsive" means patients who report that their depressive symptoms have improved through the use of citalopram but that significant depressive symptoms persist; "cannot tolerate" refers to patient report of intolerable side effects that result in a desire to discontinue the medication). Seventy-two subjects with major depressive disorder who are still symptomatic or report intolerable side effects after a 6-week open-label trial of citalopram 20mg/day ( i.e. who are not classified as responders) will be randomized to receive a higher maximum dose of citalopram (40mg/day) or switch to vilazodone during the randomization phase of the trial for 6 weeks. The hypothesis to be tested is that vilazodone will result in greater rates of treatment response and be better tolerated compared to being titrated up to a higher maximum dose (40mg/day) of citalopram. The proposed study will provide needed data on the efficacy of switching antidepressants when individuals do not fully respond to previous treatment or have intolerable side effects with a generic SSRI.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18-60;
2. Primary diagnosis of MDD. Diagnosis of MDD will be made with the Structured Clinical Interview for DSM-IV
3. Score of at least 23 on the Montgomery-Åsberg Depression Rating Scale
4. Treatment with citalopram at a dose no higher than 20mg/day for no longer than 4 weeks (subjects not currently taking an antidepressant will be started on citalopram 20mg/day for the 6-week open-label phase)
5. Ability to understand and sign the consent form.

Exclusion Criteria:

1. Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination (e.g., congestive heart failure, bradyarrhythmias).
2. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
3. Subjects considered an immediate suicide risk based on the Columbia Suicide Severity rating Scale (C-SSRS)
4. Past 3-month DSM-IV substance abuse or dependence
5. Illegal substance use based on urine toxicology screening
6. Initiation of psychotherapy or behavior therapy specifically for MDD from a mental health professional within 3 months prior to study baseline
7. Initiation of any other psychotropic medication within 2 months prior to study inclusion
8. Concomitant use of any antidepressant (except low dose doxepin, amitriptyline, trazodone when used PRN as a hypnotic).
9. Concomitant use of medications that prolong the QT interval or are CYP2C19 inhibitors (e.g., cimetidine)
10. Previous treatment with vilazodone
11. Diagnosis of bipolar I or II disorder or any psychotic disorder (anxiety disorders will be allowed as long as MDD is considered the primary psychiatric disorder)
12. Cognitive impairment that interferes with the capacity to understand and self-administer medication or provide written informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2013-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Grant, MD,JD,MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Grant JE, Redden SA, Leppink EW. Double-blind switch study of vilazodone in the treatment of major depressive disorder. Int Clin Psychopharmacol. 2017 May;32(3):121-126. doi: 10.1097/YIC.0000000000000166. PMID 28177953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Enrollment number in the Protocol Section (79) conflicts with the number of participants Started in the Participant Flow module (48) because the assessment of interested was the double-blind portion of the study. Only 48 subjects were enrolled in this phase of the study, while 79 were enrolled in the preliminary open-label phase.
Pre-assignment Details: The results reported are for the double-blind phase, not the open label citalopram phase of the study.
Period: Overall Study
Arm/Group | Vilazodone | Citalopram
Started | 20 | 28
Completed | 19 | 23
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vilazodone | Citalopram | Total
Number analyzed (Participants) | 19 | 23 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 23 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (11.3) | 38.6 (11.1) | 35.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 8 | 13 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 23 | 42

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: The entire study will last 18 weeks. For the first 6 weeks, subjects will come in once every 2 weeks. For the next 4 weeks, subjects will come in once per week. For the next 6 weeks, subjects will come in once every 2 weeks. The final visit will come 2 weeks later for a total of 11 visits where the MADRS will be administered. Only the baseline and final (last observation) assessments for the outcome measure was used in determining results, thus these are the only values included.
  MADRS scores range from 0-60, with higher scores indicating a greater level of severity. No subscales were used.
Time Frame: Baseline and final MADRS scores during the double-blind phase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vilazodone | Citalopram
Number analyzed (Participants) | 19 | 23
units on a scale
  First Randomized Visit (Visit 8) | 13.9 (5.3) | 12.7 (8.4)
  Second Randomized Visit (Visit 9) | 14.5 (4.4) | 13.2 (8.5)
  Third Randomized Visit (Visit 10) | 13.9 (5.1) | 13.5 (8.5)
  Fourth Randomized Visit (Visit 11) | 13.9 (5.3) | 12.7 (8.4)
Statistical Analysis 1: Comparison: Vilazodone vs Citalopram; Test type: Other — Linear repeated measures regression models were constructed to assess trends over time between groups where the dependent variable was outcome measure (MADRS score) and independent variables included visit, treatment group, visit by treatment group interaction, and any baseline variables that were significant between groups; p = 0.342, Regression, Linear — P-value for linear regression assessing outcome measure (MADRS score) and treatment group

ADVERSE EVENTS:
Time Frame: The adverse events reported were during the double-blind phase of the study
Arm/Group | Vilazodone | Citalopram
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 3/19 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vilazodone (N=19) | Citalopram (N=23)
Nausea (Gastrointestinal disorders) | 0 | 1
Dry Mouth (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Sexual side effects (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The sample size was likely too small to make comments about predictors of outcome and generally the study was under-powered, which would make differences difficult to detect. The study design enrolled only non-responders into the double-blind phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes